CLINICAL TRIAL: NCT05394649
Title: Intravascular Lithotripsy in Comparison to Rotational Atherectomy: An Evaluation by OFDI
Acronym: ICARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Clinique Pasteur Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2021 HONTON
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Intravascular Lithotripsy; Rotational Atherectomy; OFDI
MeSH Terms: interventions — Atherectomy, Coronary

STUDY DESIGN:
Intervention Model Description: Two parallel arms:
  * Intravascular lithotripsy arm
  * Rotational Atherectomy arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular lithotripsy arm (Experimental): Preparation of calcified lesions by intravascular lithotripsy before stenting
  Interventions: Device: Intravascular Lithotripsy
- Rotational Atherectomy arm (Active Comparator): Preparation of calcified lesions by rotational atherectomy before stenting
  Interventions: Device: Rotational Atherectomy

INTERVENTIONS:
Device: Intravascular Lithotripsy — A new device has been designed by Shockwave Medical Inc. for the treatment of calcified vascular lesions to support stent delivery: the "C2 Shockwave Medical® (IVL), Inc. coronary lithotripsy system". The system is based on lithotripsy to induce microfractures in the calcified plaque before low-pressure balloon dilation. The C2 Shockwave Medical® coronary lithotripsy (IVL) system consists of an IVL Catheter with two lithotripsy emitters enclosed within an integrated balloon, an IVL Generator, and an IVL Connector Cable.
  Arms: Intravascular lithotripsy arm
Device: Rotational Atherectomy — Rotational Atherectomy is a technique of calcic coronary plaque preparation based on the debulking of superficial calcium by a high-speed burr in order to improve vessel compliance and immediate vessel lumen gain before stenting.
  Arms: Rotational Atherectomy arm

SUMMARY:
The ICARE trial will aim to assess the efficacy of rotational atherectomy by Rotablator and Intravascular Lithotripsy by C2 Shockwave Medical® (IVL) in a randomized fashion in highly calcified lesions measured by final minimal stent area (MSA) on Optical Frequency Domain Imaging (OFDI). The investigator hypothesize that there will be no significant difference in final MSA in OFDI between the two groups after angioplasty with a last generation drug eluting stent ULTIMASTER TANSEI.

DETAILED DESCRIPTION:
Calcified coronary lesions will increase in daily percutaneous coronary intervention regarding the significant epidemiological increase of factors leading to coronary calcifications, such as hypertension, aging, and diabetes. Furthermore, calcified lesions are underdiagnosed in angiography as shown by intra-coronary imaging studies (either by OCT or IVUS), which reported that significant calcium deposits might be present in 76-83% of lesions. Calcified lesions are associated with a larger amount of periprocedural complications, as well as a poorer clinical prognosis. Standard techniques to prep the calcified plaque, such as rotational or orbital atherectomy, still have low penetration and are associated with an increase in periprocedural complications without clear clinical evidence of efficacy. More recently, there has been a growing interest in intravascular lithotripsy (IVL), which appears as an appealing option with recently published data with evidence for a safe procedure but without robust data on efficacy (sample size population, debatable effectiveness endpoint…). Although the European Society of Cardiology highlights in the latest myocardial revascularization guidelines the need for lesion preparation before stent implantation on short- and long-term clinical outcomes, no specific recommendation has been given on the use of the dedicated devices to prepare the plaque, including atherectomy, which is left to the operator assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old
2. Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for Percutaneous Coronary Intervention (PCI)
3. For patients with unstable ischemic heart disease, biomarkers (troponin or CK-MB) must be less than or equal to the upper limit of the lab (URL) normal within 12 hours prior to the procedure
4. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
5. Single de novo target lesion stenosis of protected LMCA, or LAD, RCA, or LCX (or of their branches) with:

   1. Stenosis of ≥70% and <100%
   2. or Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80
6. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm
7. The lesion length must not exceed 40 mm
8. The target vessel must have TIMI flow 3 at baseline
9. Evidence of calcification at the lesion with a B or C Mintz classification site:

   B: Moderate calcification: radiopacities are noted only during the cardiac cycle before contrast injection C: severe calcification: radiopacities are seen without cardiac motion, also before contrast injection, usually affecting both sides of the arterial lumen.
10. Ability to pass a 0.014" guidewire across the lesion
11. Ability to cross target lesion with a 2 mm balloon
12. Patient insured under the French healthcare system ("Régime National Assurance Maladie")
13. Lesions in non-target vessels requiring PCI may be treated either:

    * a. >30 days prior to the study procedure if the procedure was unsuccessful or complicated; or
    * b. >24 hours prior to the study procedure if the procedure was successful and uncomplicated (defined as a final lesion angiographic diameter stenosis <30% and TIMI 3 flow (visually assessed) for all non-target lesions and vessels without perforation, cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation, and with no post-procedure biomarker elevation >normal; or
    * c. >30 days after the study procedure d. Could be treated in the same time of the diagnosis coronarography with respect of the delay for the index procedure of the protocol as described above
14. Patient able to assess and understand the risks and benefits, to accept and participate in the study (by signing an informed consent form and knowledgeable of the information letter).
15. Patient accepting the appropriate follow-up as per study definition

Exclusion Criteria:

1. Patient age < 18 years
2. The subject is pregnant or nursing
3. Patient refusing to participate in the study or unable to give informed consent (Guardianship, curatorship or judicial safeguard)
4. Any comorbidity or condition which may reduce compliance with this protocol, including follow-up visits
5. The protected subject according to the current legislation (articles L.1121-5 to L.1121-8 of the French Code of Public Health).
6. The subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device), unless it is authorized by the concomitant study protocol.
7. Unable to tolerate dual antiplatelet therapy (i.e., aspirin, and either clopidogrel, prasugrel, or ticagrelor) for at least 6 months
8. The subject has an allergy to imaging contrast media which cannot be adequately pre-medicated
9. The subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure, defined as a clinical syndrome consistent with an acute coronary syndrome with troponin or CK-MB greater than 1 time the local laboratory's upper normal limit
10. New York Heart Association (NYHA) class III or IV heart failure
11. History of a stroke or Transient Ischemic Attack (TIA) within 6 months, or any prior intracranial hemorrhage
12. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months
13. Uncontrolled diabetes defined as an HbA1c >10%
14. Subjects in cardiogenic shock
15. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics
16. Subjects with a life expectancy of less than 1 year
17. Non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA, or PFO occlusion…) within 30 days prior to the index procedure
18. Planned non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion...)
19. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
20. High SYNTAX Score (≥33) if assessed as a standard of care, unless the local heart team has met and recommends PCI is the most appropriate treatment for the patient
21. Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel
22. Evidence of aneurysm in target vessel within 10 mm of the target Lesion
23. Unprotected left main
24. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
25. Angiographic evidence of dissection in the target vessel at baseline or after guidewire passage
26. Ejection fraction less than 30 % evaluated in TTE, angiography or MRI
27. Patient suffering of lymphoma, leukemia and other malignancies
28. Patient suffering of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
acute Minimal Stent Area (MSA) defined as in-stent minimal cross-sectional area as assessed by OFDI without In-Hospital MACE (Major Adverse Cardiac Event). | Day 1
  To assess the efficacy of IVL in a randomized fashion comparing to Rotational atherectomy by final Minimal Stent Area (MSA) measurements with Optical Frequency Domain Imaging (OFDI).

SECONDARY OUTCOMES:
MACE: Cardiac Death, all Myocardial Infarction and Target Lesion Revascularization | Day 30
  To assess safety of IVL in a randomized fashion comparing to Rotational atherectomy by checking the apparition of Major Adverse Cardiac Event (MACE) after 30 days: Cardiac death, all Myocardial Infarction (MI) and Target Lesion Revascularization (TLR)

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Groupe SAnté Victor Pauchet, Amiens
  - Clinique Rhône Durance, Avignon
  - CHU Jean Minjoz, Besançon
  - CHU Bordeaux, Bordeaux
  - Clinique Saint Augustin, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - GH Mutualiste Grenoble, Grenoble
  - Institut Cardiologique Paris sud, Massy
  - Clinique du Millénaire, Montpellier
  - Clinique Pasteur, Nancy
  - Nouvelle Clinique Nantaise, Nantes
  - CHU Nîmes, Nîmes
  - Hôpital Européen de Paris GVM la Roseraie, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - Clinique Saint Hilaire, Rouen
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No